CLINICAL TRIAL: NCT01040559
Title: Chemoembolisation of Non Resectable, Non Metastatic Hepatocellular Carcinomas Combining DC Bead Microspheres Loaded With Idarubicin (Zavedos®): Phase I Trial
Brief Title: Chemoembolisation of Non Resectable, Non Metastatic Hepatocellular Carcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Professor Laurent Bedenne, Centre Hospitalier Universitaire Dijon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDASPHERE
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Idarubicin (Experimental): Dose escalation: level0 = idarubicin 5mg, level1 = idarubicin 10mg, level2 = idarubicin 15mg, level3 = idarubicin 20mg, level4 = idarubicin 25mg
  Interventions: Drug: idarubicin

INTERVENTIONS:
Drug: idarubicin — Transarterial chemoembolization (in the hepatic artery) with idarubicin 5mg or 10 mg or 15 mg or 20 mg or 25 mg injected in a solution of 2ml DC Bead (300 µm-500µm); 1 unique course
  Other Names: 4-MDR; IMI 30; IDA

SUMMARY:
The purpose of this study is to determine the maximal tolerated dose of idarubicin for chemoembolization of non resectable non metastatic hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common malignancy and the third most common cause of cancer-related death worldwide. Most of the patients are diagnosed at intermediate-advanced stage when the sole standard treatment is transarterial chemoembolization (TACE). In the literature, survival rates in TACE studies vary widely and finally, there is no suggestion for the best chemotherapeutic agent or the optimal treatment regimen.

We hypothesise that the use of idarubicin (the most cytotoxic drug on HCC cell lines) in DC Bead would enhance the efficacy of TACE. The primary objective of the study is to determine the maximal tolerated dose of idarubicin in DC Bead for chemoembolization of non resectable non metastatic hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma cytologically or histologically proved or diagnosed according the criteria of the American Association for the Study of Liver Diseases(AASLD 2005)
* Three nodules maximum (unilobar disease without limitation in the number of nodules; 3 maximum nodules if bilobar disease [satellite nodules <1cm not included in the total sum])
* Child-Pugh score A or B7
* ECOG Performance Status < 2
* Platelet count > 50,000/µl and absolute neutrophil count (ANC) >1,000/µl
* Serum creatinine < 150 µmol/l
* Resting ejection fraction > 50% (echocardiography or isotopic method)
* Age > 18 years
* Signed written informed consent

Exclusion Criteria:

* Patients eligible for surgical resection or hepatic transplantation or radiofrequency ablation
* Extrahepatic metastases
* Known gastrointestinal bleeding up to 30 days before study entry
* Patients with anticoagulant treatment
* Evidence of portal vein thrombosis
* Pregnancy
* Clinically serious infection
* Known hypersensitivity to anthracyclines
* Known hypersensitivity to contrast medium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity assessed according NCI CTC AE v3.0 | Within the first month after chemoembolization

SECONDARY OUTCOMES:
Objective responses according criteria of the European Association for the Study of the Liver and according RECIST criteria. | 2 months
Quality of life (EORTC QLQ-C30) | 2 months
Pharmacokinetics parameters of idarubicin and idarubicinol | Within 72 hours after chemioembolization

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BEDENNE, MD Ph.D, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (1):
- Centre Hospitalier Universitaire de DIJON, Dijon, Burgundy, France

REFERENCES:
- [Derived] Anota A, Boulin M, Dabakuyo-Yonli S, Hillon P, Cercueil JP, Minello A, Jouve JL, Paoletti X, Bedenne L, Guiu B, Bonnetain F. An explorative study to assess the association between health-related quality of life and the recommended phase II dose in a phase I trial: idarubicin-loaded beads for chemoembolisation of hepatocellular carcinoma. BMJ Open. 2016 Jun 24;6(6):e010696. doi: 10.1136/bmjopen-2015-010696. PMID 27342239
- [Derived] Boulin M, Hillon P, Cercueil JP, Bonnetain F, Dabakuyo S, Minello A, Jouve JL, Lepage C, Bardou M, Wendremaire M, Guerard P, Denys A, Grandvuillemin A, Chauffert B, Bedenne L, Guiu B. Idarubicin-loaded beads for chemoembolisation of hepatocellular carcinoma: results of the IDASPHERE phase I trial. Aliment Pharmacol Ther. 2014 Jun;39(11):1301-13. doi: 10.1111/apt.12746. Epub 2014 Apr 16. PMID 24738629